CLINICAL TRIAL: NCT04273789
Title: Effect of Far Infrared Reflecting Sleepwear on Recovery and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FIRsleepwear
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Exercise Induced Muscle Damage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Prior to the study participants are informed about the study protocol, measurements and risks, but not about the study purpose. Debriefing is conducted verbally, as well as in written form and includes the signing of a second consent form.
  The experimenters conducting the measurements and analysis is not aware of the randomization. Unblinding is planned for interim analysis after 10 datasets have been collected and at study end.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- far infrared reflecting sleepwear (Experimental): Sleepwear (shorts + tshirt) with far infrared reflecting ceramic print produced by Dagsmejan AG (Zurich, Switzerland)
  Interventions: Device: Far infrared reflecting sleepwear
- Placebo sleepwear (Placebo Comparator): Sleepwear (shorts + tshirt)
  Interventions: Device: Placebo sleepwear

INTERVENTIONS:
Device: Far infrared reflecting sleepwear — 100% microlyocell sleepwear (shorts + shirt) with a ceramic print that reflects far infrared light (FIR, 5.6-1000 µm) emitted by the human body. Since FIR active garments are not powered, but reflect recycle light energy emitted by the body of the wearer, they have irradiances between 0.1-5 mW/cm^2.
  Arms: far infrared reflecting sleepwear
Device: Placebo sleepwear — 100% microlyocell sleepwear (shorts + shirt)
  Arms: Placebo sleepwear

SUMMARY:
Far infrared light (FIR, 5.6-1000 µm) penetrates our skin and reaches the underlying tissue up to 4 cm and promotes widening of the blood vessels (vasodilation). This results in increased blood flow in the tissue under the skin, without heating up the skin itself. Increased blood flow allows more oxygen to reach the muscles and more metabolic waste products to be transported away from the muscles. Studies assessing clothing containing an FDA approved ceramic particles covered yarn that reflect FIR light showed delayed onset muscle pain decreased and a reduction in inflammatory markers in professional athletes.

The aim of this study is to investigate the effect of far infrared reflecting sleepwear on night-time recovery and Sleep in a broader population, namely physically active adults (non-professional).

DETAILED DESCRIPTION:
Far infrared light (FIR, 5.6-1000 µm) penetrates our skin and reaches the underlying tissue up to 4 cm and promotes widening of the blood vessels (vasodilation). This results in increased blood flow in the tissue under the skin, without heating up the skin itself. Increased blood flow allows more oxygen to reach the muscles and more metabolic waste products to be transported away from the muscles. Thus, exposure to FIR might aid the process of recovery in muscle groups lying close to the skin.

Indeed several research groups could show that exposure to FIR aids recovery. 30 min intense far infrared exposure enhanced recovery from exercise-induced muscle damage in highly trained runners. Studies assessing clothing containing an FDA approved ceramic particles covered yarn that reflect FIR light showed delayed onset muscle pain decreased and a reduction in inflammatory markers.

Since a large part of our recovery takes place during sleep it is of interest to assess the effect of FIR on night-time recovery and sleep itself. One study showed that FIR exposure during sleep increased the amount of non-rem sleep in rats. This effect has not been replicated in humans, possibly because increased temperature is not beneficial for sleep and thus should be kept constant. The aim of this study is to investigate the effect of far infrared reflecting sleepwear on night-time recovery and sleep.

Sleepwear of a breathing and thermoregulating material, with a layer of FIR reflecting minerals printed on the outer surface, will be assessed. Physically active males are invited to participate in two bouts of exercise in the lab, separated by one week. The exercise bout targets one leg, the second week the other leg is exercised. Starting the protocol with the dominant/non-dominant leg (determined in first session) will be randomized. Participants will then wear the FIR reflecting sleepwear and placebo sleepwear respectively at home for the 7 nights following each bout of exercise.

To assess sleep quality activity will be measured using wrist worn activity trackers. To assess recovery physical performance will be measured (max. single leg force and jump height), knee range of motion and thigh circumference of each leg at before each exercise bout, after each exercise bout and at three days after each exercise bout. Per exercise bout muscle soreness will be induced in one leg of the two legs respectively, to account for a repeated bout effect.

It is hypothesized that more overnight recovery takes place during nights with FIR reflecting sleepwear compared to nights with placebo sleepwear.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (>3h of sports per week)
* BMI < 25

Exclusion Criteria:

* Sleep problems (assessed using standardized questionnaire included in entrance questionnaire)
* Cardiovascular problems (self-reported in entrance questionnaire)
* Sensitive skin/allergies that present on a skin level (self-reported in entrance questionnaire)
* Knee pain while exercising (self-reported in entrance questionnaire)
* Night shift work during study period

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Change in time of flight during jump (s) | 72 hours post exercise bout in week 1 and week 2
  Time of flight during jump is the time between offset and landing. The influence of the intervention is determined by comparing the values 72h post exercise bout of each week.
Change in maximum isometic leg force (N) | 72 hours post exercise bout in week 1 and week 2
  Maximum isometic leg force will be measured while participants are lying on their back with knees 90 Degrees bend. They press against a vertically mounted force plate. The average of 3 measurements separated by 1 minute break is used.The influence of the intervention is determined by comparing the values 72h post exercise bout of each week.
Change in leg circumference (m) | 72 hours post exercise bout in week 1 and week 2
  Circumference of the tight while standing will be measured using a measurement tape. The average of 3 measurements separated by 1 minute break is used. The influence of the intervention is determined by comparing the values 72h post exercise bout of each week.
Change in knee range of motion (Degrees) | 72 hours post exercise bout in week 1 and week 2
  Active range of motion of the knee while lying on the stomach is determined using a goniometer. The influence of the intervention is determined by comparing the values 72h post exercise bout of each week.
Change in muscle soreness (rating on visual analog scale) | 1, 2, 3, 4, 5, 6 days post exercise bout in week 1 and week 2
  Subjectively experienced delayed onset muscle soreness measured using a visual analog scale. The change in soreness over time is of interest, as well as the influence of the intervention. The influence of the intervention is determined by comparing the values 1, 2, 3, 4, 5, 6 and 7 post exercise bout of both weeks.

SECONDARY OUTCOMES:
Activity during night | 1, 2, 3, 4, 5, 6 days post exercise bout in week 1 and week 2
  Activity during night is measured using a wristworn actigraphy tracker. Based on this data sleep onset latency, sleep eficiency, sleep duration, number and duration of awakenings are calculated using validated algorithms. The influence of the intervention is determined by comparing the values 1, 2, 3, 4, 5, 6 and 7 post exercise bout of both weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, Prof. Dr., Principal Investigator — Swiss FIT
Locations (1):
- SMS lab, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
We consider uploading the actigraphy measurements to the ETH Research Collection database to make them available to other investigators.
Time Frame: The data will be ulpoaded to the research collection after study completion and is available there for a period of 15 years.
Access Criteria: Open Access
URL: https://www.research-collection.ethz.ch/